CLINICAL TRIAL: NCT05132296
Title: Mobile-Health Delivery of Lifestyle Interventions for Women With Breast Cancer Multicenter Pilot Trial
Brief Title: Mobile-Health Delivery of Lifestyle Interventions for Women With Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1190; NCI-2021-08961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1190 (Other: M D Anderson Cancer Center); UG1CA189824 (NIH)
Record Dates: First submitted 2021-09-17; First posted 2021-11-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Behavior Therapy; Practice Guidelines as Topic; Standard of Care; Nutrition Assessment; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I (CLIP) (Experimental): Patients undergo 60 minute sessions of nutrition education for 12 weeks and behavioral intervention 26 weeks. Patients receive FitBit and undergo physical activity for 30-60 minutes 5 days a week (aerobic activity) and 2 days a week (resistance training).
  Interventions: Behavioral: Behavioral Intervention; Device: FitBit; Behavioral: Nutrition Education; Other: Physical Activity; Other: Questionnaire Administration
- GROUP II (usual care) (Active Comparator): Patients have access to all usual care supportive services.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Undergo behavioral counseling
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: GROUP I (CLIP)
Other: Best Practice — Receive usual care supportive services
  Other Names: standard of care; standard therapy
  Arms: GROUP II (usual care)
Device: FitBit — Receive FitBit
  Arms: GROUP I (CLIP)
Behavioral: Nutrition Education — Receive nutrition education
  Arms: GROUP I (CLIP)
Other: Physical Activity — Undergo physical activity
  Arms: GROUP I (CLIP)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial aims to develop a lifestyle program to improve clinical outcomes in women with breast cancer who do not have a healthy diet, regular exercise habits, or ways to manage their stress well. The program will include support and counseling in healthy eating, physical activity, stress management and mindfulness, learning sleep hygiene techniques, and behavioral counseling in addition to social support. Developing a lifestyle program may help improve quality of life and encourage healthy lifestyle choices among patients diagnosed with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the feasibility of delivering a mobile, standardized, comprehensive lifestyle program in women with breast cancer (BCa).

SECONDARY OBJECTIVES:

I. Determine whether the comprehensive lifestyle intervention program (CLIP) group has reduction in body mass index (BMI) and percent body fat and weight over time.

II. Determine whether the CLIP group has improved outcomes in anthropometric measures, dietary patterns, and fitness measures and patient-reported outcomes including quality of life (QOL), fatigue, sleep disturbances, mental health, social support, and mindfulness.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients undergo 60 minute sessions of nutrition education for 12 weeks and behavioral intervention 26 weeks. Patients receive FitBit and undergo physical activity for 30-60 minutes 5 days a week (aerobic activity) and 2 days a week (resistance training).

GROUP II: Patients have access to all usual care supportive services.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage I-III BCa scheduled to undergo radiation therapy (RT) or within the first 12 months of having completed primary treatment (they do not need to have undergone RT)
* Underwent chemotherapy and surgery
* Able to read, write, and speak English
* BMI of 25 or higher
* 18 years of age or older
* Oriented to person, place, and time
* Participants must meet at least two of the following criteria related to their lifestyle at the time of diagnosis:

  * Consume less than 3 servings of fruit and vegetable/day
  * Engage in less than 75 minutes of moderate/vigorous intensity activity per week, defined as anything that causes small increases in breathing or heart rate for a sustained amount of time (e.g., brisk walking, bicycling)
  * Engage in a mind-body practice less than 4 times a month
* Access to internet connection
* Access to a tablet, laptop or computer
* Able to come to University of Texas (UT) MD Anderson or Wake Forest for blood collection
* Able to perform light physical activity. if any medical issues exist or arise that may limit performing physical activity, a medical release will be required

Exclusion Criteria:

* Have not completed chemotherapy; have a recurrent BCa diagnosis; another primary cancer diagnosis within past 5 years (not including non-melanoma skin cancers)
* Any major thought disorder (e.g., schizophrenia, dementia)
* Any major communication barriers that would preclude being able to complete the intervention (e.g., visually or hearing impaired)
* Poorly or uncontrolled diabetes in the opinion of the physician(s)
* Extreme mobility issues (e.g., unable to get in and out of a chair unassisted)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of delivering a mobile, standardized, comprehensive lifestyle program in women with BCa. | up to 9 months after study baseline
  The feasibility criteria will include consent rate (how many patients are consented in a period of time), adherence rate ( how many patients adhere to the program and finish it), and study retention rate ( how many patients that are consented stay with the program until the end/ low number of participants withdrawing from the study after consent).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT05132296/ICF_000.pdf